CLINICAL TRIAL: NCT04638686
Title: Efficacy and Safety of Dolutegravir + Lamivudine in Antiretroviral Treatment-naive Adults With HIV-1 Infection in a Multicenter Real-life Cohort Study
Brief Title: REal-Life Cohort With DOlutegravir + LAmivudina
Acronym: REDOLA
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Other Study IDs: IFJD-DOL-20-01
Record Dates: First submitted 2020-10-25; First posted 2020-11-20 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — dolutegravir; Lamivudine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Dolutegravir 50 MG — The subjects started their antiretroviral treatment containing dolutegravir once a day.
Drug: Lamivudine 300 MG — The subjects started their antiretroviral treatment containing lamivudine once a day

SUMMARY:
Since 1996, HAART based on 3-drug regimens (3DR) in people living with HIV (PLHIV) has decreased mortality and today, PLHIV have a life expectancy close to that of the general population. In the last decade new drugs have improved tolerance and posology of these treatment. However PLHIV needs to continue the treatment and will likely remain on antiviral therapy for many years. In the recent period, active research is being sought with the aim of improving the dosage and reducing the amount of drugs necessary to maintain efficacy, to avoid the possible cumulative effects of long-term antiretroviral therapy (ART). Two-drug regimens (2DRs) have been investigated as a means for reducing the number of antiretroviral agents (ARVs) taken by individuals who need lifelong ART. Dovato® (Dolutegravir/lamivudine) has been evaluated in two phase III studies (GEMINI-1 and GEMINI-2) in treatment-naive adults achieving non inferiority according to the US Food and Drug Administration (FDA) Snapshot algorithm. These data led to the approval of the fixed-dose combination of dolutegravir/lamivudine as a once-daily, single-tablet 2DR by the FDA and the European Medicines Agency. Actual update to the US Department of Health and Human Services treatment guidelines for HIV-1 infection and European AIDS Clinical Society guidelines indicate Dovato ® as an initial treatment in HIV-naÏve patients. However there is no real- life cohort data. Our aim is to provide information related to effectiveness and tolerability/safety in naïve patients when used in routine clinical practice. It has been already published results from the phase III study in pretreatment adult patients.

Our results in real life have encouraged us to conduct a multicenter cohort study in patients who have already started their first antiretroviral therapy with dolutegravir (DTG) + lamivudine (3TC), to verify efficacy and tolerance in real life. Our hypothesis is that the data will be similar to those reported in clinical trials.

DETAILED DESCRIPTION:
Our primary objective of this study is to analyze the proportion of individuals (HIV naïve patients) who has initiated 3TC (300 mg p.o. q 24 h) plus DTG (50 mg p.o. q 24 h), and who achieve viral suppression (HIV-1 RNA ≤50 copies/mL) at weeks 48.

Secondary objectives are: to analyze the proportion of individuals who achieve viral suppression (HIV-1 RNA ≤50 copies/mL) at weeks 24 and 96, to describe absolute values and changes from ART initiation in CD4+ cells count and CD4:CD8 ratio at 24, 48 and 96 weeks, Changes from ART initiation in creatinine clearance anda fasting lipids at weeks 24, 48 and 96, and the proportion of subjects who discontinue treatment and reasons for discontinuations

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age diagnosed with HIV.
* Naïve antiretroviral treatment with dolutegravir/lamivudine initiated between July 2018 and March 2020.
* Patients who agree to participate and sign the informed consent form of the study
* Patients lost to follow up or died prior to the inclusion in the study (Ethics Committee agreement for exemption from obtaining informed consent in these cases).

Exclusion Criteria:

* Patient < 18 years of age.
* Patients who don't agree to participate and don't sign the informed consent.
* Current pregnancy or breastfeeding.
* No effective contraception for FRP women.
* Evidence of DTG or 3TC resistance genotype*
* Hepatitis B (HBV) infection
* Severe hepatic impairment or unstable liver disease
* Moderate to severe renal impairment
* AIDS defining illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is an open, multicenter and prospective cohort of HIV-infected adult patients who have initiated Dolutegravir/lamivudine as first line treatment for HIV-1 infection prior to be included in study. We hope to include 200 patients. Patient management will be according to the standard of care.
  We will collect data related to efficacy, tolerance, and discontinuations due any reasons (lost to follow-up, withdrawal of consent, switching,..).
  We will carry out an analysis by intention to treat according to the snapshot criteria defined by the FDA ±12 weeks window in the context of routine clinical practice (±2 weeks in w-4 analysis), considering as virological failure those patients who discontinue the treatment for any reason, loss to follow-up, withdraw informed consent or those who die for causes unrelated to the treatment
Sampling Method: Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of individuals who achieve viral suppression (HIV-1 RNA ≤50 copies/mL) at weeks 48 | 48 weeks
  HIV-1 RNA ≤50 copies/mL at 48 weeks

SECONDARY OUTCOMES:
Proportion of individuals who achieve viral suppression (HIV-1 RNA ≤50 copies/mL) at weeks 24 and 96 | weeks 24 and 96
  HIV-1 RNA ≤50 copies/mL at 24 and 96 weeks
Absolute values and changes from ART initiation in CD4+ cells count at 24, 48 and 96 weeks | weeks 24, 48 and 96
  CD4 (cel/μL) at weeks 0, 24,48 and 96
Absolute values and changes from ART initiation in CD4:CD8 ratio at 24, 48 and 96 | weeks 24, 48 and 96
  CD4/CD8 (ratio) at weeks 0, 24,48 and 96
Changes from ART initiation in creatinine clearance at weeks 24, 48 and 96. | weeks 24, 48 and 96
  creatinine clearance (mg/dL) at weeks 0, 24, 48 and 96.
Changes from ART initiation in fasting lipids (total cholesterol, HDL cholesterol, LDL) cholesterol, triglycerides and ratio of total cholesterol to HDL cholesterol) at weeks 24, 48 and 96 | weeks 24, 48 and 96
  total cholesterol, HDL cholesterol, LDL (mg/dL) at weeks 0, 24, 48 and 96.
Proportion of subjects who discontinue treatment and reasons for discontinuations | weeks 48 and 96
  number of subjects who discontinue treatment and reasons for these discontinuations

CONTACTS AND LOCATIONS:
Locations (1):
- Alfonso Cabello, Madrid, Spain

REFERENCES:
- [Background] Cahn P, Madero JS, Arribas JR, Antinori A, Ortiz R, Clarke AE, Hung CC, Rockstroh JK, Girard PM, Sievers J, Man C, Currie A, Underwood M, Tenorio AR, Pappa K, Wynne B, Fettiplace A, Gartland M, Aboud M, Smith K; GEMINI Study Team. Dolutegravir plus lamivudine versus dolutegravir plus tenofovir disoproxil fumarate and emtricitabine in antiretroviral-naive adults with HIV-1 infection (GEMINI-1 and GEMINI-2): week 48 results from two multicentre, double-blind, randomised, non-inferiority, phase 3 trials. Lancet. 2019 Jan 12;393(10167):143-155. doi: 10.1016/S0140-6736(18)32462-0. Epub 2018 Nov 9. PMID 30420123
- [Background] Radford M, Parks DC, Ferrante S, Punekar Y. Comparative efficacy and safety and dolutegravir and lamivudine in treatment naive HIV patients. AIDS. 2019 Sep 1;33(11):1739-1749. doi: 10.1097/QAD.0000000000002285. PMID 31180906
- [Background] van Wyk J, Ajana F, Bisshop F, De Wit S, Osiyemi O, Portilla Sogorb J, Routy JP, Wyen C, Ait-Khaled M, Nascimento MC, Pappa KA, Wang R, Wright J, Tenorio AR, Wynne B, Aboud M, Gartland MJ, Smith KY. Efficacy and Safety of Switching to Dolutegravir/Lamivudine Fixed-Dose 2-Drug Regimen vs Continuing a Tenofovir Alafenamide-Based 3- or 4-Drug Regimen for Maintenance of Virologic Suppression in Adults Living With Human Immunodeficiency Virus Type 1: Phase 3, Randomized, Noninferiority TANGO Study. Clin Infect Dis. 2020 Nov 5;71(8):1920-1929. doi: 10.1093/cid/ciz1243. PMID 31905383
- [Background] Taiwo BO, Marconi VC, Berzins B, Moser CB, Nyaku AN, Fichtenbaum CJ, Benson CA, Wilkin T, Koletar SL, Colasanti J, Acosta EP, Li JZ, Sax PE. Dolutegravir Plus Lamivudine Maintains Human Immunodeficiency Virus-1 Suppression Through Week 48 in a Pilot Randomized Trial. Clin Infect Dis. 2018 May 17;66(11):1794-1797. doi: 10.1093/cid/cix1131. PMID 29293895
- [Background] Joly V, Burdet C, Landman R, Vigan M, Charpentier C, Katlama C, Cabie A, Benalycherif A, Peytavin G, Yeni P, Mentre F, Argoud AL, Amri I, Descamps D, Yazdanpanah Y; LAMIDOL Study Group. Dolutegravir and lamivudine maintenance therapy in HIV-1 virologically suppressed patients: results of the ANRS 167 trial (LAMIDOL). J Antimicrob Chemother. 2019 Mar 1;74(3):739-745. doi: 10.1093/jac/dky467. PMID 30476165
- [Derived] Cabello-Ubeda A, Lopez Bernardo de Quiros JC, Mena A, Torralba M, Martin Carbonero L, Gutierrez A, Vergas J, Pinto A, Tejerina F, Palmier E, Sanz J, Gorgolas M, Pulido F. Dolutegravir (DTG) + Lamivudine (3 TC) in Antiretroviral-Naive Adults With HIV With and Without Genotypic Resistance Testing Results: 96-Week Effectiveness and Tolerability of REDOLA Study. J Acquir Immune Defic Syndr. 2025 Oct 1;100(2):e4-e7. doi: 10.1097/QAI.0000000000003721. No abstract available. PMID 40673705